CLINICAL TRIAL: NCT05393375
Title: Arthrogryposis Multiplex Congenita in Pediatric Age: Correlation Between MUScular MRI and Functional Evaluation
Acronym: AMUSE
Status: Completed | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-AMUSE
Record Dates: First submitted 2022-05-17; First posted 2022-05-26 (Actual); Last update posted 2023-01-04 (Actual); Status verified 2022-05

CONDITIONS: Arthrogryposis Multiplex Congenita; AMC-Arthrogryposis Multiplex Congenita; Pediatric ALL
Keywords: Arthrogryposis Multiplex Congenita; Pediatric; Mercuri Score; MRI; Fibro-adipous infiltration; Functional capacity; Rehabilitation; Retrospective observational study
MeSH Terms: conditions — Arthrogryposis; Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group 1 Amyoplasia: Patients with diagnosis of Amyoplasia
  Interventions: Other: No intervention
- Group 2 Distal Arthrogryposis: Patients with diagnosis of Distal Arthrogryposis
  Interventions: Other: No intervention
- Group 3 Other: Patients with diagnosis of other form of AMC
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
The aim of our study is to evaluate the correlation between quantified fibro-adipous infiltration of muscles on MRI assessed by MERCURI Score and the functional abilities (deficiencies, activity limitations and social participation of pediatric patients with arthrogryposis.

DETAILED DESCRIPTION:
Arthrogryposis multiplex congenita (AMC) is a group of rare diseases characterized by joint contractures at two or more distinct joint levels at birth. More than 400 causes are currently known. The prevalence is estimated at 1/3000 to 1/2000. Joint limitations are not progressive, but the functional consequences have a lifelong impact on patients.

Correlations between fibro-adipous infiltration and muscular deficits have already been studied in other neuromuscular diseases such as Pompe disease or Duchenne muscular dystrophy. These studies concluded on a good correlation between disease progression and severity, muscle strength, and fatty infiltration assessed by Mercuri score. The investigators concluded that muscular MRI can be used as a non-invasive biomarker and a tool to follow the progression of neuromuscular disease and help evaluate the potential effects of therapies.

The aim of this project is to define whether MRI could also be used as a tool, through the assessment of muscle fatty infiltration, to help predict the functional abilities of our patients with AMC, and more specifically the two most frequent types, Amyoplasia and distal arthrogryposis.

The investigators will analyze fatty infiltration measured by muscle MRI and quantify it using the MERCURI score which was developed by Mercuri et al. (Mercuri et al. 2002) as a semi-quantitative score to quantify fibro-adipose muscle infiltration on muscle MRI.

The investigators will evaluate musculoskeletal deficiencies and limitations of activity from data obtained from patients followed in our AMC reference center at the University Hospital Grenoble Alpes (CHUGA).

The investigators will include data from 220 children, 97 of whom have had a complete check-up including a muscle MRI. The investigators will study the existence of a correlation between this score and the deficiencies and limitations of activity.

The investigators will then evaluate the potential predictive role of fatty infiltration measured on MRI in the functional abilities of the patients.

This characterization will help to better determine and anticipate the functional capacities of our patients from the beginning of their treatment to improve their functional prognosis.

This initial work could enhance the reflection on the biomechanical modeling of joints and key functions such as standing and the acquisition of walking, in order to pave the way for rehabilitation and compensation methods that are better adapted to patient's needs.

ELIGIBILITY:
Inclusion Criteria:

* age < 18 at the first clinical evaluation or follow up exclusively in CHUGA pediatric rehabilitation unit
* Clinical or molecular diagnosis of AMC established by geneticists at CHUGA
* functional evaluation during consultation and follow-up in CHUGA pediatric rehabilitation unit
* Muscle MRI of upper limbs, lower limbs and trunk performed at CHUGA pediatric radiology unit

Exclusion Criteria:

* Contra indication MRI.
* MRI non exploitable.
* Patient under guardianship or deprived of liberty

Ages: 0 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatric patient from PARART registry (Paediatric and Adult Registry on ARThrogryposis) evaluated in the reference center (RC) for Arthrogryposis Multiplex Congenita from 2010 until 2021). All patients were evaluated by a geneticist, and had a complete check up in the pediatric PMR unit (physical medicine and rehabilitation physician, physiotherapists, occupational and speech therapists) and had imaging analysis by whole body muscular MRI.
Sampling Method: Non-Probability Sample
Enrollment: 97 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-11-01 (Actual)

PRIMARY OUTCOMES:
Mercuri Scores of upper limbs, trunk, and lower limbs evaluated on muscle MRI T1 | through study completion, an average of 1 year
  The degree of fatty muscle infiltration was assessed on muscular MRI and quantified by Mercuri score, each muscle was staged as follows:
  1. Normal appearance, 2. Mild involvement (30-60% fatty infiltration). 3. Moderate involvement (>60% fatty infiltration). 4. Severe involvement (complete infiltration).
  The degree of muscle fat infiltration was assessed with at least 2 visible slices, and performed by two independent operators. In case of divergent assessments, a consensus was reached after discussion.

SECONDARY OUTCOMES:
Muscular weakness | through study completion, an average of 1 year
  Muscular weakness assessed by function (flexion, extension etc.) and not by each muscle, using the Medical Research Council (MRC) scale (from 0 to 5).
  The quotation was as follows: 0, no contraction; 1, flicker or trace of contraction; 2, active movement possible only with gravity eliminated; 3, active movement against gravity in the whole range of motion; 4, active movement against gravity and resistance; 5, quasi-normal strength) Evaluated by physiotherapists, occupational therapists and physician during evaluation.
Passive range of motion (PROM) | through study completion, an average of 1 year
  Evaluated by physiotherapists; the range of motion of each movement in degrees was normalized with respect to the normal maximal movement, expressed as percentages
Reaching score | through study completion, an average of 1 year
  Reaching capacity was assessed by ad hoc test. Patients were instructed to successively touch some body targets with upper limbs : mouth, head, forehead, neck, back, stomach, gluteal region, opposite shoulders, ipsilateral shoulders, knee, feet, "Beggar's pose", "position of the oath", and "Zenith Pose". Each gesture was marked "yes" if successful or "no" if not.
  Responses were transformed into a binary variable with "yes" being worth 1 and "no" being worth 0 to allow for statistical correlations afterwards. The total score was calculated on both sides averaged and ranged from 0 to 14 points
Ambulatory status | through study completion, an average of 1 year
  Ambulatory statuses were gathered by the teams during the check-ups as well as the age of acquisition of walking if available and the use or not of technical aids
School status | through study completion, an average of 1 year
  Type of schooling (mainstream education, adapted schooling, presence of a carer)
Activity limitation | through study completion, an average of 1 year
  Gathered evaluating living habits and essential acts of daily life such as element of the Functional Independence Measure (FIM) : feeding, dressing, potty training, toileting, schooling, transfers, locomotion, and also existence of leisure, hobby, presence of human or technical helps.
Surgery History | through study completion, an average of 1 year
  Surgical history for each patient
Human and technical Help | through study completion, an average of 1 year
  use of a technical aid (manual or electric wheelchair ...), or humain for daily life activities

CONTACTS AND LOCATIONS:
Overall Officials: Klaus DIETERICH, MD, Study Director — CHU Grenoble Alpes
Locations (1):
- CHU Grenoble Alpes, La Tronche, France

REFERENCES:
- [Result] Hall JG. Arthrogryposis multiplex congenita: etiology, genetics, classification, diagnostic approach, and general aspects. J Pediatr Orthop B. 1997 Jul;6(3):159-66. PMID 9260643
- [Result] Mercuri E, Pichiecchio A, Counsell S, Allsop J, Cini C, Jungbluth H, Uggetti C, Bydder G. A short protocol for muscle MRI in children with muscular dystrophies. Eur J Paediatr Neurol. 2002;6(6):305-7. doi: 10.1016/s1090-3798(02)90617-3. PMID 12401454
- [Result] Figueroa-Bonaparte S, Segovia S, Llauger J, Belmonte I, Pedrosa I, Alejaldre A, Mayos M, Suarez-Cuartin G, Gallardo E, Illa I, Diaz-Manera J; Spanish Pompe Study Group. Muscle MRI Findings in Childhood/Adult Onset Pompe Disease Correlate with Muscle Function. PLoS One. 2016 Oct 6;11(10):e0163493. doi: 10.1371/journal.pone.0163493. eCollection 2016. PMID 27711114
- [Result] Quijano-Roy S, Avila-Smirnow D, Carlier RY; WB-MRI muscle study group. Whole body muscle MRI protocol: pattern recognition in early onset NM disorders. Neuromuscul Disord. 2012 Oct 1;22 Suppl 2:S68-84. doi: 10.1016/j.nmd.2012.08.003. PMID 22980770
- [Result] Dieterich K, Le Tanno P, Kimber E, Jouk PS, Hall J, Giampietro P. The diagnostic workup in a patient with AMC: Overview of the clinical evaluation and paraclinical analyses with review of the literature. Am J Med Genet C Semin Med Genet. 2019 Sep;181(3):337-344. doi: 10.1002/ajmg.c.31730. Epub 2019 Aug 1. PMID 31368648